CLINICAL TRIAL: NCT01746017
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Oral Doses of LY2922470 in Healthy Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2922470 in Healthy Participants and Participants With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14796; I6K-FW-GLEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2922470

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Part A) (Placebo Comparator): Single oral dose of placebo administered to healthy participants in up to 1 of 4 study periods in Part A
  Interventions: Drug: Placebo
- LY2922470 (Part A) (Experimental): Single ascending dose of LY2922470 [starting at 1 milligram (mg)] administered orally to healthy participants in up to 3 of 4 study periods in Part A
  Interventions: Drug: LY2922470
- Placebo (Part B) (Placebo Comparator): Single oral dose of placebo administered to participants with type 2 diabetes mellitus (T2DM) in up to 1 of 3 study periods in Part B
  Interventions: Drug: Placebo
- LY2922470 (Part B) (Experimental): Single ascending dose of LY2922470 administered orally to participants with T2DM in up to 2 of 3 study periods in Part B. Dose determined by Part A
  Interventions: Drug: LY2922470

INTERVENTIONS:
Drug: Placebo — Administered orally as capsules
  Arms: Placebo (Part A); Placebo (Part B)
Drug: LY2922470 — Administered orally as capsules
  Arms: LY2922470 (Part A); LY2922470 (Part B)

SUMMARY:
The aim of this trial is to evaluate the safety of the study drug in healthy participant and participant with diabetes. It will investigate how much of the study drug gets into the blood stream and how long it takes the body to get rid of it. Information about any side effects that may occur will also be collected.

The study consists of two parts. Part A will study healthy participants in up to 4 dosing periods over approximately 6 weeks. Part B will study participants with diabetes in up to 3 dosing periods over approximately 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Must be a male, or a female who cannot become pregnant, and who is either a healthy participant, or who has type 2 diabetes
* Have a screening body mass index (BMI) of at least 18.0 kilograms per square meter (kg/m^2)
* Have blood pressure, pulse rate, blood and urine laboratory test results acceptable for the study

For participants with Type 2 Diabetes Mellitus (T2DM):

* Do not have any change to their diabetes treatment (exercise with or without metformin) for at least 4 weeks prior to screening.
* Have a glycated hemoglobin (HbA1c) value of greater than or equal to 6% and less than or equal to 11% at screening

Exclusion Criteria:

For all participants:

* Are currently participating in another clinical study or completed one in the last 30 days
* Are allergic to LY2922470 or other related drugs
* Have a history of significant heart, lung, liver, kidney, stomach or brain disease, or have any medical problems which may cause an increased risk during the study
* Have electrocardiogram (ECG) readings that are not suitable for the study
* Are infected with hepatitis B
* Are infected with human immunodeficiency virus (HIV)
* Have donated more than 450 milliliter (mL) of blood in the last 3 months or if have donated any blood in the last month
* Have a regular alcohol intake greater than 21 units/week (male), or 14 units/week (female), or are unwilling to stop alcohol as required by the study restrictions (1 unit = 360 mL of beer, or 150 mL of wine, or 45 mL of spirits)
* Smoke more than 10 cigarettes per day or are not willing to abstain from smoking while at the clinic.

For participants with T2DM:

* Have had heart disease or stroke within 6 months before entering the study
* Have health complications due to poorly controlled diabetes as shown by blood and urine laboratory test results or based on physical examination and medical assessment as determined by the study doctor
* Have been hospitalized for poor control of diabetes (keto-acidotic episode) in the last 6 months
* Have used insulin to control diabetes in the last 1 year
* Show symptoms of high blood sugar, for example (e.g.), frequent urination, always feeling thirsty, or unexpected weight loss

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 2-part dose escalation study: Part A in healthy participants and Part B in participants with type 2 diabetes mellitus (T2DM). Participants in Part A participated in up to 4 intervention periods and participants in Part B participated in up to 3 intervention periods. There was an at least 8 days washout interval between each dosing.
Groups:
- Part A Cohort 1 Sequence 1: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: Placebo; Period 2: 10 milligrams (mg) LY2922470; Period 3: 90mg LY2922470; Period 4: 540mg LY2922470;
- Part A Cohort 1 Sequence 2: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 1mg LY2922470; Period 2: 10mg LY2922470; Period 3: 90mg LY2922470; Period 4: Placebo;
- Part A Cohort 1 Sequence 3: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 1mg LY2922470; Period 2: Placebo; Period 3: 90mg LY2922470; Period 4: 540mg LY2922470;
- Part A Cohort 1 Sequence 4: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 1mg LY2922470; Period 2: 90mg LY2922470; Period 3: Placebo; Period 4: 540mg LY2922470;
- Part A Cohort 2 Sequence 1: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 3mg LY2922470; Period 2: 30mg LY2922470; Period 3: Placebo; Period 4: 1350mg LY2922470;
- Part A Cohort 2 Sequence 2: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 3mg LY2922470; Period 2: 30mg LY2922470; Period 3: 270mg LY2922470; Period 4: Placebo;
- Part A Cohort 2 Sequence 3: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 3mg LY2922470; Period 2: Placebo; Period 3: 270mg LY2922470; Period 4: 1350mg LY2922470;
- Part A Cohort 2 Sequence 4: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: Placebo; Period 2: 30mg LY2922470; Period 3: 270mg LY2922470; Period 4: 1350mg LY2922470;
- Part B Sequence 1: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: Placebo; Period 2: 540mg LY2922470; Period 3: 1080mg LY2922470;
- Part B Sequence 2: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 270mg LY2922470; Period 2: 540mg LY2922470; Period 3: Placebo;
- Part B Sequence 3: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 270mg LY2922470; Period 2: Placebo; Period 3: 1080mg LY2922470;
Period: Period 1
Arm/Group | Part A Cohort 1 Sequence 1 | Part A Cohort 1 Sequence 2 | Part A Cohort 1 Sequence 3 | Part A Cohort 1 Sequence 4 | Part A Cohort 2 Sequence 1 | Part A Cohort 2 Sequence 2 | Part A Cohort 2 Sequence 3 | Part A Cohort 2 Sequence 4 | Part B Sequence 1 | Part B Sequence 2 | Part B Sequence 3
Started | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3
Received at Least 1 Dose of Study Drug | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part A Cohort 1 Sequence 1 | Part A Cohort 1 Sequence 2 | Part A Cohort 1 Sequence 3 | Part A Cohort 1 Sequence 4 | Part A Cohort 2 Sequence 1 | Part A Cohort 2 Sequence 2 | Part A Cohort 2 Sequence 3 | Part A Cohort 2 Sequence 4 | Part B Sequence 1 | Part B Sequence 2 | Part B Sequence 3
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A Cohort 1 Sequence 1 | Part A Cohort 1 Sequence 2 | Part A Cohort 1 Sequence 3 | Part A Cohort 1 Sequence 4 | Part A Cohort 2 Sequence 1 | Part A Cohort 2 Sequence 2 | Part A Cohort 2 Sequence 3 | Part A Cohort 2 Sequence 4 | Part B Sequence 1 | Part B Sequence 2 | Part B Sequence 3
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Part A Cohort 1 Sequence 1 | Part A Cohort 1 Sequence 2 | Part A Cohort 1 Sequence 3 | Part A Cohort 1 Sequence 4 | Part A Cohort 2 Sequence 1 | Part A Cohort 2 Sequence 2 | Part A Cohort 2 Sequence 3 | Part A Cohort 2 Sequence 4 | Part B Sequence 1 | Part B Sequence 2 | Part B Sequence 3
Started | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 0 (Part B occurred only for 3 periods.) | 0 (Part B occurred only for 3 periods.) | 0 (Part B occurred only for 3 periods.)
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Part A Cohort 1 Sequence 4: Participants received either Placebo or LY2922470 capsules orally as per the below dosing sequence in each period.
  Period 1: 1mg LY2922470; Period 2: 10mg LY2922470; Period 3: Placebo; Period 4: 540mg LY2922470;
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1 Sequence 1 | Part A Cohort 1 Sequence 2 | Part A Cohort 1 Sequence 3 | Part A Cohort 1 Sequence 4 | Part A Cohort 2 Sequence 1 | Part A Cohort 2 Sequence 2 | Part A Cohort 2 Sequence 3 | Part A Cohort 2 Sequence 4 | Part B Sequence 1 | Part B Sequence 2 | Part B Sequence 3 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 26
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion up to 33 days
Population: All enrolled participants who received at least 1 dose of study drug. Participants were analyzed based on the treatment they received.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Part A): Single oral dose of placebo administered to healthy participants in 1 of 4 study periods.
- 1 mg (Part A): Single oral dose of 1 mg LY2922470 administered to healthy participants in 1 of 4 study periods.
- 3 mg (Part A): Single oral dose of 3 mg LY2922470 administered to healthy participants in 1 of 4 study periods.
- 10 mg (Part A): Single oral dose of 10 mg LY2922470 administered to healthy participants in 1 of 4 study periods.
- 30 mg (Part A): Single oral dose of 30 mg LY2922470 administered to healthy participants in 1 of 4 study periods.
- 90 mg (Part A): Single oral dose of 90 mg LY2922470 administered to healthy participants in 1 of 4 study periods.
- 270 mg (Part A): Single oral dose of 270 mg LY2922470 administered to healthy participants in 1 of 4 study periods.
- 540 mg (Part A): Single oral dose of 540 mg LY2922470 administered to healthy participants in 1 of 4 study periods.
- 1350 mg (Part A): Single oral dose of 1350 mg LY2922470 administered to healthy participants in 1 of 4 study periods.
- Placebo (Part B): Single oral dose of placebo administered to participants with T2DM in 1 of 3 study periods.
- 270 mg (Part B): Single oral dose of 270 mg LY2922470 administered to participants with T2DM in 1 of 3 study periods.
- 540 mg (Part B): Single oral dose of 540 mg LY2922470 administered to participants with T2DM in 1 of 3 study periods.
- 1080 mg (Part B): Single oral dose of 1080 mg LY2922470 administered to participants with T2DM in 1 of 3 study periods.
Arm/Group | Placebo (Part A) | 1 mg (Part A) | 3 mg (Part A) | 10 mg (Part A) | 30 mg (Part A) | 90 mg (Part A) | 270 mg (Part A) | 540 mg (Part A) | 1350 mg (Part A) | Placebo (Part B) | 270 mg (Part B) | 540 mg (Part B) | 1080 mg (Part B)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve of LY2922470 From Time Zero to 24 Hours [AUC(0-24)]
Time Frame: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 18, 24, 48, 96 and 192 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug and had sufficient pharmacokinetics data to calculate AUC(0-24). Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | 1 mg (Part A) | 3 mg (Part A) | 10 mg (Part A) | 30 mg (Part A) | 90 mg (Part A) | 270 mg (Part A) | 540 mg (Part A) | 1350 mg (Part A) | 270 mg (Part B) | 540 mg (Part B) | 1080 mg (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
nanograms*hour/milliliter (ng*hr/mL) | 52.1 (30) | 194 (26) | 658 (33) | 2340 (24) | 6110 (20) | 13300 (31) | 23900 (50) | 50200 (46) | 15200 (31) | 33700 (30) | 78200 (42)

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2922470
Time Frame: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 18, 24, 48, 96 and 192 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug and had sufficient pharmacokinetics data to calculate Cmax. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 1 mg (Part A) | 3 mg (Part A) | 10 mg (Part A) | 30 mg (Part A) | 90 mg (Part A) | 270 mg (Part A) | 540 mg (Part A) | 1350 mg (Part A) | 270 mg (Part B) | 540 mg (Part B) | 1080 mg (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
nanograms/milliliter (ng/mL) | 11.1 (15) | 30.5 (33) | 111 (37) | 457 (38) | 1030 (33) | 2320 (21) | 4130 (37) | 6050 (50) | 2000 (37) | 3780 (56) | 7950 (30)

4. Secondary Outcome: Change From Baseline in Blood Glucose Area Under the Effective Concentration Curve From Time Zero to 24 Hours [AUEC(0-24)]
Description: Least Squares (LS) mean values were adjusted for baseline, treatment, period, treatment sequence, participant and error.
Time Frame: Baseline (predose for Part A and Day -1 time-matched for Part B), 24 hours postdose
Population: All participants who received at least 1 dose of study drug with both baseline and 24 hours postdose glucose AUEC(0-24) values. Participants were analyzed based on the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: millimoles*hour/Liter (mmol*h/L)
Arm/Group | Placebo (Part A) | 1 mg (Part A) | 3 mg (Part A) | 10 mg (Part A) | 30 mg (Part A) | 90 mg (Part A) | 270 mg (Part A) | 540 mg (Part A) | 1350 mg (Part A) | Placebo (Part B) | 270 mg (Part B) | 540 mg (Part B) | 1080 mg (Part B)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
millimoles*hour/Liter (mmol*h/L) | 6.88 (1.52) | 10.49 (3.64) | 1.29 (3.67) | 8.20 (3.46) | 2.04 (3.43) | 3.68 (3.47) | 10.76 (3.37) | -0.34 (3.46) | 7.34 (3.61) | -11.47 (3.68) | -19.95 (9.08) | -21.01 (9.10) | -27.19 (9.07)

5. Secondary Outcome: Change From Baseline in C-Peptide Area Under the Effective Concentration Curve From Time Zero to 6 Hours [AUEC(0-6)]
Description: LS mean values were adjusted for baseline, treatment, period, treatment sequence, participant and error.
Time Frame: Baseline (predose for Part A and Day -1 time-matched for Part B), 6 hours postdose
Population: All participants who received at least 1 dose of study drug with both baseline and 6 hours postdose C-peptide AUEC(0-6) values. Participants were analyzed based on the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: picomoles*hour/Liter (pmol*h/L)
Arm/Group | Placebo (Part A) | 1 mg (Part A) | 3 mg (Part A) | 10 mg (Part A) | 30 mg (Part A) | 90 mg (Part A) | 270 mg (Part A) | 540 mg (Part A) | 1350 mg (Part A) | Placebo (Part B) | 270 mg (Part B) | 540 mg (Part B) | 1080 mg (Part B)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
picomoles*hour/Liter (pmol*h/L) | 7349.88 (871.01) | 6314.08 (1257.47) | 6270.86 (1262.57) | 5465.01 (1257.11) | 6351.84 (1242.12) | 6651.32 (1264.87) | 7472.28 (1259.71) | 6499.90 (1263.96) | 6442.33 (1307.48) | 1518.13 (560.25) | 1657.94 (1428.92) | 5496.32 (1430.24) | 1790.26 (1428.57)

ADVERSE EVENTS:
Arm/Group | Placebo (Part A) | 1 mg (Part A) | 3 mg (Part A) | 10 mg (Part A) | 30 mg (Part A) | 90 mg (Part A) | 270 mg (Part A) | 540 mg (Part A) | 1350 mg (Part A) | Placebo (Part B) | 270 mg (Part B) | 540 mg (Part B) | 1080 mg (Part B)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/15 | 1/6 | 1/6 | 2/6 | 3/6 | 3/6 | 3/6 | 1/6 | 2/6 | 3/9 | 3/6 | 2/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=15) | 1 mg (Part A) (N=6) | 3 mg (Part A) (N=6) | 10 mg (Part A) (N=6) | 30 mg (Part A) (N=6) | 90 mg (Part A) (N=6) | 270 mg (Part A) (N=6) | 540 mg (Part A) (N=6) | 1350 mg (Part A) (N=6) | Placebo (Part B) (N=9) | 270 mg (Part B) (N=6) | 540 mg (Part B) (N=6) | 1080 mg (Part B) (N=6)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes